CLINICAL TRIAL: NCT06985108
Title: Comparison of Nasal Endotracheal Tube and Spiral Tube for Nasotracheal Intubation in Pediatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dicle University (Other)
Responsible Party: Principal Investigator, Zülfü SAVAŞ, medicine doctor anesthesiology specialist, Dicle University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 171/2025
Record Dates: First submitted 2025-05-06; First posted 2025-05-22 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Epistaxis
Keywords: nazotracheal intubation; north polar tube; epistaxis; spiral tube
MeSH Terms: conditions — Epistaxis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- north polar tube (Active Comparator): patients who intubated with north polar tube
  Interventions: Procedure: nazotracheal intubation
- spiral tube (Active Comparator): patients who intubated with spiral tube
  Interventions: Procedure: nazotracheal intubation

INTERVENTIONS:
Procedure: nazotracheal intubation — intubation tube will be placed from nasal orifice through nazopharyngeal pathway to place into trachea

SUMMARY:
Nasotracheal intubation is often preferred in patients under general anesthesia for maxillofacial surgery or dental treatment to ensure airway safety and to work more comfortably in the surgical field. Compared to orotracheal intubation, the nasotracheal approach is a more convenient option, especially during procedures whose surgical site is in the oral region.

Standard spiral intubation tubes are commonly used for nasotracheal intubation. However, there are also pre-shaped nasal intubation tubes that are specially designed to better fit the nasopharyngeal anatomical structure. The North Polar Tube, one of the most prominent of these tubes, is preferred because it is easier to insert through the nasal route and reduces potential trauma.

In our hospital, nasal intubation is routinely preferred in pediatric patients under general anesthesia for dental procedures. However, there are not enough comparative studies in the literature on the advantages and disadvantages of different intubation tubes used in these applications, especially in the pediatric age group.

In our hospital, nasal intubation is routinely performed in pediatric patients undergoing general anesthesia for dental treatments. In this study, the investigators will compare the spiral intubation tube and nasotracheal intubation tube used for intubation of these patients in terms of epistaxis, intubation time and difficulty of intubation.

DETAILED DESCRIPTION:
During our study, 96 patients between the ages of 3-18 years with appropriate criteria between 01.05.2025-01.08.2025 will be recruited for general anesthesia.

Patients will be taken to the operating room and after routine monitoring methods (SpO2, Pulse, Non invasive blood pressure) are used and data are recorded, 1 mg/kg midazolam, 1 mg/kg lidocaine, 2 mcg/kg fentanyl, 2-3 mg/kg propofol and 0.6-1.2 mg/kg rocuronium will be administered intravenously. Before intubation, patients will be randomly distributed into groups by closed envelope method (Group 1: NPT, Group 2: Spiral Tube) and intubation will be performed using nasal intubation tube or spiral tube. The procedures performed are daily routine procedures and no new procedure will be performed on the patient.

Vital measurements at the 1st and 5th minutes after intubation will be recorded. Anesthesia maintenance will be provided with 2-3% sevoflurane 50% oxygen 50% air mixture.

After intubation, the presence and severity of epistaxis, if any; presence of intra-oral bleeding, use of Magill forceps, duration of intubation, difficulty of intubation (number of intubation attempts, need for video laryngoscope use), whether laryngeal compression (Sellick maneuver) was applied and glottic degree (Cormack-Lehane classification) data will be recorded. When nasotracheal intubation cannot be performed, orotracheal intubation will be performed and patients will be excluded from the study.

Inclusion Criteria; Being between 3-18 years old

* No anomaly preventing nasal intubation
* To be in ASA1-2 classification according to ASA criteria

Exclusion Criteria;

* Lack of consent of the patient/ relatives
* Facial anomaly that prevents nasal intubation
* Being in the ASA3-4 group according to ASA criteria

ELIGIBILITY:
Inclusion Criteria:

* Being between 3-18 years old
* No anomaly preventing nasal intubation
* To be in ASA1-2 classification according to ASA criteria

Exclusion Criteria:

* Lack of consent of the patient/ relatives
* Facial anomaly that prevents nasal intubation
* Being in the ASA3-4 group according to ASA criteria

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 98 (Actual)
Dates: Start 2025-05-02 (Actual); Primary Completion 2025-08-30 (Actual); Study Completion 2025-10-30 (Actual)

PRIMARY OUTCOMES:
epistaxis frequency | perioperative period
  epistaxis presence will be controlled at 0. minute and 5. minute after intubation. Epistaxis occurancy will be noted as present/absent. More incidence of epistaxis will be related to worse outcome.
severity of epistaxis | perioperative period
  epistaxis severity will be measured at 0.and 5. minute after intubation. Severity will be classified as; none:no blood observed on either the surface of the tube or the posterior pharyngeal wall mild:blood apparent on the surface of the tube or posterior pharyngeal wall moderate: pooling of blood on the posterior pharyngeal wall severe: large amount of blood in the pharynx impeding nasotracheal intubation and necessitating urgent orotracheal intubation The outcome gets worse as it goes from none to severe.

SECONDARY OUTCOMES:
intubation duration | perioperative
  intubation duration will be noted in seconds and there is predicted minimum and maximum values. Prolonged intubation time is related to worse outcome.
intubation difficulty | perioperative
  To assessment of intubation difficulty; number of attempts, Cormack lehane score, usage of Magill forceps, usage of Video laryngoscope and need to Sellick maneuver will be noted.
  Higher number of attempts will indicate worse outcome. Other evaluations will be in a yes/no format. İf the yes rate be higher than the no rate outcome will be accepted as worse

CONTACTS AND LOCATIONS:
Overall Officials: Fikret Salik, specialist, Study Director — Dicle university faculty of medicine
Locations (1):
- Dicle university Faculty of dentistry, Diyarbakır, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
all collected IDP
Supporting Information: Study Protocol
Time Frame: 3 months after publication of results
Access Criteria: medicine doctors, dentists

REFERENCES:
- See also: Latest publication about similar work-up — https://pubmed.ncbi.nlm.nih.gov/38548948/

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-05-06): https://cdn.clinicaltrials.gov/large-docs/08/NCT06985108/Prot_SAP_ICF_000.pdf